CLINICAL TRIAL: NCT06101121
Title: Performance and Safety of Lubri-cream for Pain Minimization During Urethral Catheterization and Cystoscopy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: B. Braun Medical SA (Industry)
Responsible Party: Sponsor
Other Study IDs: HC-O-H-2113
Record Dates: First submitted 2023-10-20; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Urethral Catheter; Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Urethral catherisation: Observation time will start with placement of catheter and will end with catheter removal or if any complication appears, whatever occurs first. In this case, the observational time will be 1 day when a bladder catheterization is undergone.
  Interventions: Device: Lubri-Cream
- Cytoscopy: Observation time will start with placement of catheter and will end with catheter removal or if any complication appears, whatever occurs first. In this case, the observational time will be the time which the catheterization lasts.
  Interventions: Device: Lubri-Cream

INTERVENTIONS:
Device: Lubri-Cream — Lubri-cream is indicated as a surface lubricant for bladder catheterization and cystoscopy. It will be slowly applied on the device, exerting gentle and constant pressure on the tube. Its contents will be evenly distrubuted from the tip to a suitable distance according to the technique to be performed. An individualized dose will be applied according to the technique to be performed and at the discretion of the healthcare professional

SUMMARY:
The primary aim of this study is to collect clinical data on the performance of Lubri-cream applied in routine clinical practice.

Safety and efficacy parameters of Lubri-cream in lubrication on bladder catheterization and cystoscopy will be assessed.

DETAILED DESCRIPTION:
The study is designed as a prospective, multicenter, single-group, observational study to evaluate Lubri-cream for urethral catheterization and cystoscopies lubrication. At least 2 different centers located in Spain will participate.

It is primarily aimed to collect data on the performance of the product under investigation in a large patient population when used in routine clinical practice. Safety and performance of Lubri-cream will be assessed to study the pain minimization when patients undergo urethral catheterization and cystoscopy procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Any patient who needs urethral catheterization or cystoscopy (rigid or flexible).
* Signed informed consent

Exclusion Criteria:

* Contraindications as stated in the Instructions for Use
* Any medical or psychological disorder that, in the investigator's opinion, may interfere with the patient's ability to give informed consent and comply with the study procedures
* Inclusion in another investigational study in the field of urethral catheterization or cystoscopy which could interfere with the clinical practice regarding the application and care of the Investigational Product.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: See eligibility criteria
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Performance of Lubri-cream based on the pain minimization when patients undergo urethral catheterization and cystoscopy procedures. | During catheter insertion, catheter removal and if any complication appears (AE/SAEs)
  Patients' perception of pain level will be measured using the VAS, a visual scale of 10 cm in length, anchored by word descriptors at each end where "0 cm" means "no pain" and "10 cm" means "worst ever pain". The "zero-end" will be marked with "no pain" and the "10 cm"-end will be marked as "worst ever pain".

SECONDARY OUTCOMES:
Safety of Lubri-cream based on routinely measured clinical parameters | During catheter insertion and catheter removal
  Occurrence of adverse events after its use in patients

CONTACTS AND LOCATIONS:
Overall Officials: Anna Maria Martínez, Dr., Principal Investigator — Hospital Universitari Mútua Terrassa

IPD SHARING:
Plan to Share IPD: Undecided